CLINICAL TRIAL: NCT05353426
Title: Paragastric Lesser Omentum Neural Block to Prevent Visceral Pain After Laparoscopic Sleeve Gastrectomy: A Randomized Clinical Trial Protocol.
Brief Title: Paragastric Autonomic Blockade to Prevent Visceral Pain After Laparoscopic Sleeve Gastrectomy
Acronym: PG-ANB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Simón Bolívar (Other)
Responsible Party: Principal Investigator, Yaneth Herazo Beltran, Designated Investigator, Universidad Simón Bolívar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO-CEI-USB-CE-0394-00
Record Dates: First submitted 2022-04-16; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Visceral Pain; Bariatric Surgery Candidate; Pain, Postoperative; Vomiting, Postoperative; Nausea, Postoperative
Keywords: Paragastric; Autonomic Block; Visceral pain; Opioids; Multimodal pain
MeSH Terms: conditions — Visceral Pain; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomized clinical trial involving patients undergoing laparoscopic sleeve gastrectomy.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PG-ANB Block (Experimental): The paragastric lesser omentum neural block is performed with a 25-gauge needle attached to a venous catheter extension introduced through the left 12-mm port. The needle is capped during its introduction, and the cap is removed inside the abdomen using a grasper and kept under direct vision. Infiltration of 20 mL of non-diluted 0.5% bupivacaine is performed at six levels with careful aspiration preceding fluid infiltration. Four of the areas are next to the vagus nerves and branches, and two are in the vicinity of the common hepatic and left gastric arteries
  Interventions: Procedure: Paragastric autonomic neural blockade
- Control (No Intervention): No paragastric neural block is performed in the control group. The same standard analgesic protocol consisting of acetaminophen (1 g) and morphine (3-5 mg) is used in all patients before extubation and TAP block is performed in both groups (control and experimental)

INTERVENTIONS:
Procedure: Paragastric autonomic neural blockade — Paragastric autonomic neural blockade with Bupivacaine
  Other Names: Laparoscopic transverses abdomens plane (TAP) block (To Both the control and experimental arms); Laparoscopic sleeve gastrectomy(LSG) to all patients
  Arms: PG-ANB Block

SUMMARY:
Visceral pain (VP) following laparoscopic sleeve gastrectomy remains a substantial problem. VP is associated with autonomic symptoms, especially nausea and vomiting, and is unresponsive to traditional pain management algorithms aimed at alleviating somatic (incisional) pain. The present study was performed to evaluate the safety and effectiveness of laparoscopic paragastric autonomic neural blockade (PG-ANB) in managing the symptoms associated with VP following sleeve gastrectomy.

DETAILED DESCRIPTION:
Introduction Although seldom discussed, visceral pain (VP) is the most significant source of pain in the first 24 hours following laparoscopic sleeve gastrectomy (LSG) and other laparoscopic procedures (1). The somatic pain induced by surgical trauma to the abdominal wall after LSG is effectively managed using conventional analgesia and transversus abdominis plane (TAP) blocks (2-4). In contrast, the visceral, colicky pain patients experience after LSG does not respond well to traditional pain management regimens. During the last 15 years at our institutions, we have used many analgesic strategies to manage these burdensome symptoms in more than 2000 LSG procedures. Despite these efforts, no analgesic strategies have been satisfactorily effective (5,8,9).

Autonomic nerve blocks have been described in the pain management literature. Specifically, celiac ganglia blocks have been reported in managing chronic pain caused by foregut malignancies or pancreatitis (11,12). In these patients, neuraxial blocks have been demonstrated to be safe and effective methods of chronic pain management. To our knowledge, however, paragastric autonomic neural blockade (PG-ANB) has not been performed as part of perioperative multimodal pain management algorithms in gastrointestinal surgery. The two proposed main mechanisms of action of this autonomic blockade are a reduction in the parasympathetic influence over the stomach, which reverses its increased muscular tone and deactivates mechanosensitive receptors in the organ wall, and blockade of the afferent sympathetic fibers that convey VP to the spinal cord (13).

In a pilot observational study involving 35 patients, we observed improvement in the severity of VP in the epigastric and retrosternal areas as well as improvement in associated autonomic symptoms following PG-ANB (14). The effect was most pronounced during the immediate postoperative period but persisted until discharge. Analgesic requirements and the presence of nausea and vomiting were also reduced. The current study was performed to further validate these preliminary findings through a randomized, double-blinded controlled trial.

Study design This prospective, double-blinded, randomized clinical trial involved patients undergoing laparoscopic sleeve gastrectomy at two high-volume institutions. The patients were randomized to laparoscopic transversus abdominis plane block with or without PG-ANB.

Sample size Previously published data have indicated that differences of 1 to 2 points on an 11-point visual analog pain scale are clinically significant (15-17). Based on these prior studies, we chose a difference of 1 point as the minimum clinically significant difference for sample size calculation and assumed a standard deviation of 2 points. With a p-value of 0.05 and a power of 0.80, we estimated that a total of 128 patients would need to be enrolled in this study. To allow for any potential loss to follow-up, we enrolled 150 patients in the study.

Randomization and blinding Randomization was performed using sealed envelopes prepared by the data manager and stratified by institution in blocks of six. The data manager stored the randomization list containing the final treatment assignments. Only the data manager had access to the randomization list throughout the study. These sealed envelopes were placed in the patients' charts and could not be opened until the patient was in the operating room under general anesthesia. At that point, the surgeon became cognizant of the procedure to perform but did not participate in assessing the patient or collecting data. Both the patient and the investigator assessing the patient were blinded to the treatment arm assignments. The investigator evaluated the patients for vital signs, pain scores, autonomic symptoms, and analgesic requirements and recorded the information.

Data collection The patients' age, sex, body mass index, current medications, and medical and surgical history were prospectively recorded at the preoperative clinic visit during study enrollment with informed consent. An analog pain scale survey was administered by an investigator blinded to the patients' groups at 1 hour postoperatively (in the recovery room), 8 hours postoperatively, and the following morning. The investigator recorded the need for analgesics; the presence of nausea, vomiting, retching, excessive salivation, hiccups; and vital signs.

Statistical analysis Continuous outcome variables were compared with two-sample t-tests. Categorical and binary outcome variables were compared using chi-squared tests. Patient-reported pain scores were further compared using linear regression with the surgeon who operated and the location of the procedure as covariates to assess the effect of the surgeon and location on the primary outcome.

Postoperative recovery protocol All patients received proton pump inhibitors, conventional antiemetics, and a scheduled baseline analgesic such as acetaminophen (1 g intravenously every 6 hours) or dipyrone (1 g intravenously every 6 hours). The first-line rescue analgesic was a nonsteroidal anti-inflammatory drug such as diclofenac (intravenously every 12 hours) together with hyoscine butylbromide (0.2 mg intravenously every 12 hours), and the second-line rescue analgesic was tramadol (1 mg per ideal body weight intravenously every 6 hours). Tramadol was the only opioid derivative used. A popsicle was offered the afternoon after surgery, and clear fluids were started the following day. Patients were discharged from the hospital at noon the day after surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who were scheduled for LSG at each participating institution from 25 August 2021 to 8 February 2022 and consented to study participation.

Exclusion Criteria:

* the exclusion criteria were an age of <18 years.
* the performance of concomitant procedures in addition to LSG.
* allergies to medications included in the postoperative management protocol.
* anesthetic complications related to the LSG that would alter the postoperative management protocol.
* surgical complications related to the LSG that would alter the postoperative management protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
The patient-reported pain scores using an 11-point visual analog scale for pain( 11 being the worse pain). | Outcomes were assessed up to 24 hours after surgery during the period of inpatient admission following LSG.
  An analog pain scale survey was administered by an investigator blinded to the patients' groups at 1 hour postoperatively (in the recovery room), 8 hours postoperatively, and the following morning

SECONDARY OUTCOMES:
The secondary outcomes were analgesic requirements. | The recorded administered doses of analgesics were assessed up 24 hours after surgery during the period of inpatient admission following LSG.
  The investigator recorded the need for additional doses of the analgesics, established in the protocol, at one, eight and twenty four hours after surgery.
The secondary outcome was present of nauseas | Recorded up to 24 hours after surgery
  The investigator recorded the present of nausea at 1, 8 and 24 hours after surgery.
The secondary outcome was present of vomiting | Recorded up to 24 hours after surgery
  The investigator recorded the present of vomiting at 1, 8 and 24 hours after surgery.
The secondary outcome was present of retching | Recorded up to 24 hours after surgery
  The investigator recorded the present of retching at 1, 8 and 24 hours after surgery.
The secondary outcome was present of excessive salivation | Recorded up to 24 hours after surgery
  The investigator recorded the present of excessive salivation at 1, 8 and 24 hours after surgery.
The secondary outcome was present of hiccups | Recorded up to 24 hours after surgery
  The investigator recorded the present of hiccups at 1, 8 and 24 hours after surgery.
The secondary outcomes was the mean arterial blood pressure | Recorded at 10 minutes after blockade
  The investigator recorded the mean arterial blood pressure 10 minutes after blockade.
The secondary outcomes was the median heart rate | Recorded at 10 minutes after blockade.
  The investigator recorded the median heart rate 10 minutes after blockade.
The secondary outcomes was the mean arterial blood pressure. | Recorded up to 24 hours after surgery
  The investigator recorded the mean arterial blood pressure at 1, 8 and 24 hours after surgery.
The secondary outcomes was the median heart rate. | Recorded up to 24 hours after surgery
  The investigator recorded the median heart rate at 1, 8 and 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Daes, MD FACS, Study Director — Academic Director Clinica portoazul, Barranquilla, Colombia
Locations (1):
- Clinica Portoazul, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daes J, Jimenez ME, Said N, Daza JC, Dennis R. Laparoscopic sleeve gastrectomy: symptoms of gastroesophageal reflux can be reduced by changes in surgical technique. Obes Surg. 2012 Dec;22(12):1874-9. doi: 10.1007/s11695-012-0746-5. PMID 22915063
- [Background] Browning KN, Travagli RA. Central nervous system control of gastrointestinal motility and secretion and modulation of gastrointestinal functions. Compr Physiol. 2014 Oct;4(4):1339-68. doi: 10.1002/cphy.c130055. PMID 25428846
- [Background] Akinci D, Akhan O. Celiac ganglia block. Eur J Radiol. 2005 Sep;55(3):355-61. doi: 10.1016/j.ejrad.2005.03.008. PMID 16129244
- [Background] Gress F, Schmitt C, Sherman S, Ikenberry S, Lehman G. A prospective randomized comparison of endoscopic ultrasound- and computed tomography-guided celiac plexus block for managing chronic pancreatitis pain. Am J Gastroenterol. 1999 Apr;94(4):900-5. doi: 10.1111/j.1572-0241.1999.01042.x. PMID 10201454
- [Background] Ruiz-Tovar J, Munoz JL, Gonzalez J, Zubiaga L, Garcia A, Jimenez M, Ferrigni C, Duran M. Postoperative pain after laparoscopic sleeve gastrectomy: comparison of three analgesic schemes (isolated intravenous analgesia, epidural analgesia associated with intravenous analgesia and port-sites infiltration with bupivacaine associated with intravenous analgesia). Surg Endosc. 2017 Jan;31(1):231-236. doi: 10.1007/s00464-016-4961-3. Epub 2016 May 13. PMID 27177956
- [Background] Iamaroon A, Tangwiwat S, Nivatpumin P, Lertwacha T, Rungmongkolsab P, Pangthipampai P. Risk Factors for Moderate to Severe Pain during the First 24 Hours after Laparoscopic Bariatric Surgery While Receiving Intravenous Patient-Controlled Analgesia. Anesthesiol Res Pract. 2019 Oct 3;2019:6593736. doi: 10.1155/2019/6593736. eCollection 2019. PMID 31687018
- [Background] Tian C, Lee Y, Oparin Y, Hong D, Shanthanna H. Benefits of Transversus Abdominis Plane Block on Postoperative Analgesia after Bariatric Surgery: A Systematic Review and Meta-Analysis. Pain Physician. 2021 Aug;24(5):345-358. PMID 34323436
- [Background] Joris J, Thiry E, Paris P, Weerts J, Lamy M. Pain after laparoscopic cholecystectomy: characteristics and effect of intraperitoneal bupivacaine. Anesth Analg. 1995 Aug;81(2):379-84. doi: 10.1097/00000539-199508000-00029. PMID 7618731
- [Result] Daes J, Pantoja R, Hanssen A, et al.Paragastric, lesser omentum neural block to prevent early visceral pain after laparoscopic sleeve gastrectomy: A randomized clinical trial protocol. Revista Colombiana de Cirugia 2022;37:27-32. https://doi.org/10.30944/20117582.1017